CLINICAL TRIAL: NCT04813224
Title: Psychological Intervention in Women Victims of Childhood Sexual Abuse: A Randomized Clinical Trial Comparing EMDR Psychotherapy and Trauma-Based Cognitive Therapy.
Brief Title: Intervention Through EMDR and CBT With Women Victim of Childhood Sexual Abuse. A Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Internacional de Valencia (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, María Teresa Mitjans Lafont, Full time psychology professor Universidad Internacional de Valencia, Universidad Internacional de Valencia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VIU-EMDR-TFCBT
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Posttraumatic Stress Disorder; Somatization; Obsessive-Compulsive Disorder; Depression; Anxiety; Hostility; Dissociative Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder; Depression; Anxiety Disorders; Dissociative Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: The patients are not aware that there is another intervention and that they will receive both of them. The participants are not related and do not know each other. The conditions of the study are only known by the researcher, the therapists, and the Committee for the Evaluation and Monitoring of Research with Human Beings of the Universidad Internacional de Valencia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAUMA CENTERED EMDR-BASED TREATMENT (Experimental): Phase 1) Client history before session 1 Phase 2) Preparation for the treatment of the traumatic event, with psycho education and regulation strategies.
  Phases 3 to 6) Gives the sense of Safety (safe place, past resource, desired future-PC, timeline) control structure, order, differentiation of past & present (move concretely between past danger to present safety) EMD strategy gives containment boundaries to current T-Episode.
  Phase 7) Session closure A group debriefing of the experience will take place, and some of the stabilization exercises Phase 8) Re-Evaluation This phase will take place immediately after the group intervention. It assesses which participants may need individual attention and which may need further evaluation to identify the nature and extent of their symptoms.
  Interventions: Behavioral: TRAUMA CENTERED EMDR-BASED TREATMENT and TRAUMA-FOCUSED CBT-BASED TREATMENT
- TRAUMA-FOCUSED CBT-BASED TREATMENT (Active Comparator): TF-CBT is an evidence-based therapeutic approach to improve symptoms of PTSD as well as affective or cognitive and behavioral problems. The treatment will consist of three phases that will include: Psychoeducation, Relaxation-Mindfulness, Emotional regulation skills, Cognitive coping skills, Narration and processing of trauma, Exposure / Desensitization of memories of the trauma, Self-esteem and future goals. The treatment is composed by 3 phases: 1) Phase 1: TF-CBT Coping Skills for Complex Traumas. Phase 2: Narration of trauma and processing of complicated trauma. Phase 3: Consolidation and closure of the treatment. Each case is delivered to the participants in a maximum of 3 sessions per phase.
  Interventions: Behavioral: TRAUMA CENTERED EMDR-BASED TREATMENT and TRAUMA-FOCUSED CBT-BASED TREATMENT

INTERVENTIONS:
Behavioral: TRAUMA CENTERED EMDR-BASED TREATMENT and TRAUMA-FOCUSED CBT-BASED TREATMENT — Psychological evidence-based intervention for the reduction of the impact of childhood sexual abuse.

SUMMARY:
This study evaluates the effectiveness of two types of therapy for the treatment of sexual abuse psychological impact on a sample of Spanish women. The participants will receive first Trauma-Focused Cognitive Behavioral Therapy and Eye Movement Desensitization and Reprocessing treatments in order to observe the impact on symptoms of Posttraumatic Stress Disorder, somatization, obsessive-compulsive symptoms, anxiety, aggressiveness and dissociate symptoms.

DETAILED DESCRIPTION:
The experience of sexual abuse in childhood is one of the forms of interpersonal victimization most associated with the development of psychological problems since it involves a serious violation of the rights and sexual and affective freedom of children and adolescents. The different types of child abuse and neglect are, in turn, associated with moderately severe psychological sequelae in adulthood. Its effects in adult life can affect physical, psychological, and social functioning and generate psychopathological alterations, being the most frequent consequences. Women who were abused in childhood, in their adult life more frequently presented sexual dysfunction and less perceived sexual satisfaction, less trust, and more difficulties in communicating with the partner.

Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) is an evidence-based treatment model designed to help patients (children, adolescents, youth) and their families overcome the symptoms resulting from exposure to a traumatic experience. Numerous investigations that support it, today it is considered a well-established intervention for the treatment of post-traumatic stress and associated symptoms.

Desensitization and reprocessing psychotherapy using eye movements. It is one of the transdiagnostic psychotherapeutic models of choice in international guidelines for dealing with the sequelae of traumatic life experiences. Trauma-focused treatment carried out with the EMDR therapeutic approach is feasible and safe for patients with PTSD derived from childhood sexual abuse.

A Randomized Clinical Trial is proposed, without a control group, and assignment to two types of treatment 1) TF -CBT, 2) EMDR.

After the initial evaluation, the participants will be randomly assigned to one of the two treatments. Subsequently, and after allowing the same time period that the intervention protocols will last, they will be evaluated again to measure changes without having received treatment. After this second evaluation, they will receive the treatment protocol to which they have been assigned after randomization. After receiving the first treatment, they will be evaluated again. After this evaluation, they will receive the other protocol of the intervention. Finally, after finishing the second intervention, they will be evaluated again. Thus, for example, participants who first received TF-CBT will subsequently receive the EMDR intervention, and participants who first received the EMDR intervention will subsequently receive the TF-CBT intervention. In this way, it will be possible to evaluate both the effectiveness of each of the protocols separately (intragroup comparison of each treatment condition), as well as the level of effectiveness obtained by comparing both treatment groups (intergroup comparison, after the application of each type of intervention ).

The subjective measures will include the following Psychometrics:

Satisfaction with life scale Rosenberg Self-Esteem Scale Symptom Checklist-90-Revised Post-Traumatic Stress Disorder Symptom Severity Scale according to DSM-5 (EGS-R) DSM-5 Personality Inventory - Short Version (PID-5-BF) Adults Scale of emotional regulation difficulties Dissociative Symptom Scale Satisfaction scale with received treatment Satisfaction scale with received treatment

ELIGIBILITY:
Inclusion Criteria:

* present symptoms related to the post-traumatic sequelae of having had an experience of sexual abuse in childhood.
* The traumatic experience is accessible to explicit memory.
* The participant has shared her experience at least in a context of containment and is able to talk about it.

Exclusion Criteria:

* Enfermedad mental grave.
* Extreme scores on both the personality questionnaire and the Psychopathology questionnaire in the indicator of global severity, paranoid ideation, and psychoticism.
* Any problem of addiction to alcohol or other substances at the time of the evaluation, etc. that may interfere with adherence to treatment and group dynamics.
* Being currently in treatment to treat the traumatic experience.
* Present severe dissociative symptoms, beyond those typical of the PTSD diagnosis.
* Extreme scores on the dissociation scale in the pathological ideation items.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The treatment will be directed only to adult women that suffered sexual child abuse, due to the characteristics possible to access the sample in an established center that only offers treatment to women. Future studies can be conducted with both genders.
Enrollment: 50 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-12-16 (Estimated); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
Decrease in the scores of the Post-Traumatic Stress Disorder Symptom Severity Scale according to the DSM-5 (EGS-R) | 4.5 months, after receiving both interventions.
  The Revised Symptom Severity Scale for Post-Traumatic Stress Disorder (PTSD) consists of 21 items, based on the DSM-5 diagnostic criteria, and is used to assess the severity of the symptoms of this clinical picture. It is a structured assessment instrument, with responses measured with a Likert-type scale from 0 to 3 according to the frequency and intensity of the symptoms.
  This scale has a nuclear part (EGS-R) and a complementary part. The core part consists of 21 central items (range: 0-63 points) in correspondence with the diagnostic criteria of the DSM-5 (APA, 2013): 5 refer to intrusion (range: 0-15), 3 to avoidance behavioral / cognitive (range: 0-9), 7 to cognitive disturbances and negative mood (AC / EAN) (range: 0-21) and 6 to hyperarousal (range: 0-18), as well as 4 additional ones referred to dissociation (range: 0-12).
  It is expected that in all these subscales they will be significantly reduced (P <0.05) scores by patients after the treatments.
Decrease in the scores of the clinical symptoms measured using the Symptom Checklist-90-Revised (SCL-R) | 4.5 months, after receiving both interventions.
  The SCL-90-R is a self-administered questionnaire that presents 90 elements that describe symptoms and requires the individual to indicate through a Likert-type scale graduated between 0 (not at all) and 4 (a lot or extremely) to what extent they have annoying feeling for each of the symptoms described.
  The questionnaire allows obtaining three global indices and 10 symptomatic dimensions: 1) Global Severity Index, 2) Total Positive Symptoms, 3) Positive Discomfort Index, 4) Somatization, 5) Obsession-compulsion, 6) Interpersonal sensitivity, 7) Depression, 8) Anxiety, 9) Hostility, 10) Phobic anxiety, 11) Paranoid ideation, 12) Psychoticism, 13) Additional scale (ADI). It collects seven symptoms that have a relevant factorial weight on different scales. A clinically significant reduction (P <0.05) is expected in the Global Severity index, in the Total of positive symptoms, in the positive index of discomfort, in depression and anxiety.
Decrease in the scores on the Dissociative Symptom Scale. | 4.5 months, after receiving both interventions.
  It is a 28-item self-administered scale, developed by Bernstein and Putnam (1986), designed to measure dissociative symptomatology. Items are scored, according to the frequency of each dissociative experience, in a range of 0 to 100, where 0 represents "never" and 100 "always." The center points represent 50% of the time. The global score is the sum of the score assigned to each item, divided by 28. The higher the global score, the more severe the dissociative symptoms, therefore improvement is indicated by a decrease in the DES score.
  A clinically significant reduction (P <0.05) in the total score of this scale is expected after the treatments.

SECONDARY OUTCOMES:
Increase in the scores of the Satisfaction with Life Scale (SWLS) | 4.5 months, after receiving both interventions.
  This instrument consists of 5 items in which the participants must indicate how much they agree with each question, with response options in Likert format from 1 (totally disagree) to 7 (totally agree) ). Scores range from a minimum of 5 to a maximum of 35, where higher scores indicate greater satisfaction with life. A clinically significant increase (P <0.05) in the global score of this scale is expected after the treatments.
Increase in the scores of the Rosenberg Self-Esteem Scale | 4.5 months, after receiving both interventions.
  This instrument assesses the feeling of satisfaction that a person has about himself. The questionnaire is made up of 10 items (half of the items are positively stated and the other half negatively) whose contents focus on the general feelings of respect and acceptance towards oneself. The items are answered in a four-point Likert format (1 = Strongly agree, 2 = Agree, 3 = Disagree, 4 = Strongly disagree) depending on the degree of agreement with the statement made. The total score ranges from 10 to 40 points, distinguishing between low self-esteem (scores less than or equal to 25), medium (from 26 to 29) and high (equal to or greater than 30).
  A clinically significant increase (P <0.05) in the global score of this scale is expected after the treatments.
Increase in the scores of the Emotional Regulation Difficulties Scale (DERS) | 4.5 months, after receiving both interventions.
  This scale assesses different aspects of the emotional regulation process in which there may be difficulties: emotional lack of control, daily interference, emotional inattention, emotional confusion and emotional rejection. The first factor, "Emotional lack of control", includes items from two scales of the original version: "Difficulty in impulse control" and "Limited access to regulation strategies". The rest of the factors correspond to the remaining subscales of the original version, although the labels were slightly modified with respect to the originals for reasons of simplification and adaptation to Spanish: "Emotional rejection", "Everyday interference", "Emotional neglect", "Emotional confusion." A clinically significant decrease (P <0.05) is expected in the scores of the factors: "Emotional lack of control", "Emotional rejection", "Daily interference", "Emotional inattention" and "Emotional confusion"

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Molero Zafra, MD, Study Chair — Universidad Internacional de Valencia; Alejandro Domínguez Rodríguez, PhD, Study Chair — Universidad Internacional de Valencia; Marian Pérez Marín, PhD, Study Chair — University of Valencia
Locations (1):
- Asociación Contra los Abusos Sexuales en la Infancia (ACASI), Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study. The protocol of the study is currently in progress to be published, in this article will be included such study protocol, the informed consent is already shared in the register of clinical trials.
Supporting Information: ICF
Time Frame: This data will be available approximately in December 2021 and it will be permanently available. It will be shared in the databases of the journal where the article(s) will be published.
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Bisson JI, Roberts NP, Andrew M, Cooper R, Lewis C. Psychological therapies for chronic post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2013 Dec 13;2013(12):CD003388. doi: 10.1002/14651858.CD003388.pub4. PMID 24338345
- [Background] Canton-Cortes D, Canton J, Cortes MR. The interactive effect of blame attribution with characteristics of child sexual abuse on posttraumatic stress disorder. J Nerv Ment Dis. 2012 Apr;200(4):329-35. doi: 10.1097/NMD.0b013e31824cc078. PMID 22456587
- [Background] Cohen JA, Mannarino AP, Kliethermes M, Murray LA. Trauma-focused CBT for youth with complex trauma. Child Abuse Negl. 2012 Jun;36(6):528-41. doi: 10.1016/j.chiabu.2012.03.007. Epub 2012 Jun 30. PMID 22749612
- [Background] Davidson PR, Parker KC. Eye movement desensitization and reprocessing (EMDR): a meta-analysis. J Consult Clin Psychol. 2001 Apr;69(2):305-16. doi: 10.1037//0022-006x.69.2.305. PMID 11393607
- [Background] De Jongh A, Groenland GN, Sanches S, Bongaerts H, Voorendonk EM, Van Minnen A. The impact of brief intensive trauma-focused treatment for PTSD on symptoms of borderline personality disorder. Eur J Psychotraumatol. 2020 Feb 14;11(1):1721142. doi: 10.1080/20008198.2020.1721142. eCollection 2020. PMID 32128048
- [Background] Deblinger E, Pollio E, Dorsey S. Applying Trauma-Focused Cognitive-Behavioral Therapy in Group Format. Child Maltreat. 2016 Feb;21(1):59-73. doi: 10.1177/1077559515620668. Epub 2015 Dec 23. PMID 26701151
- [Background] Deblinger E, Mannarino AP, Cohen JA, Runyon MK, Steer RA. Trauma-focused cognitive behavioral therapy for children: impact of the trauma narrative and treatment length. Depress Anxiety. 2011 Jan;28(1):67-75. doi: 10.1002/da.20744. Epub 2010 Sep 9. PMID 20830695
- [Background] Karadag M, Gokcen C, Sarp AS. EMDR therapy in children and adolescents who have post-traumatic stress disorder: a six-week follow-up study. Int J Psychiatry Clin Pract. 2020 Mar;24(1):77-82. doi: 10.1080/13651501.2019.1682171. Epub 2019 Oct 30. PMID 31663396
- [Background] Lee CW, Cuijpers P. A meta-analysis of the contribution of eye movements in processing emotional memories. J Behav Ther Exp Psychiatry. 2013 Jun;44(2):231-9. doi: 10.1016/j.jbtep.2012.11.001. Epub 2012 Nov 20. PMID 23266601
- [Background] Ostacoli L, Carletto S, Cavallo M, Baldomir-Gago P, Di Lorenzo G, Fernandez I, Hase M, Justo-Alonso A, Lehnung M, Migliaretti G, Oliva F, Pagani M, Recarey-Eiris S, Torta R, Tumani V, Gonzalez-Vazquez AI, Hofmann A. Comparison of Eye Movement Desensitization Reprocessing and Cognitive Behavioral Therapy as Adjunctive Treatments for Recurrent Depression: The European Depression EMDR Network (EDEN) Randomized Controlled Trial. Front Psychol. 2018 Feb 13;9:74. doi: 10.3389/fpsyg.2018.00074. eCollection 2018. PMID 29487548
- [Background] Horst F, Den Oudsten B, Zijlstra W, de Jongh A, Lobbestael J, De Vries J. Cognitive Behavioral Therapy vs. Eye Movement Desensitization and Reprocessing for Treating Panic Disorder: A Randomized Controlled Trial. Front Psychol. 2017 Aug 18;8:1409. doi: 10.3389/fpsyg.2017.01409. eCollection 2017. PMID 28868042
- [Result] Bernstein EM, Putnam FW. Development, reliability, and validity of a dissociation scale. J Nerv Ment Dis. 1986 Dec;174(12):727-35. doi: 10.1097/00005053-198612000-00004. PMID 3783140
- [Result] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Result] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Result] Elhai JD, Gray MJ, Kashdan TB, Franklin CL. Which instruments are most commonly used to assess traumatic event exposure and posttraumatic effects?: A survey of traumatic stress professionals. J Trauma Stress. 2005 Oct;18(5):541-5. doi: 10.1002/jts.20062. PMID 16281252
- [Result] Gutierrez F, Aluja A, Peri JM, Calvo N, Ferrer M, Bailles E, Gutierrez-Zotes JA, Garriz M, Caseras X, Markon KE, Krueger RF. Psychometric Properties of the Spanish PID-5 in a Clinical and a Community Sample. Assessment. 2017 Apr;24(3):326-336. doi: 10.1177/1073191115606518. Epub 2016 Jul 28. PMID 26391204
- [Derived] Molero-Zafra M, Fernandez-Garcia O, Mitjans-Lafont MT, Perez-Marin M, Hernandez-Jimenez MJ. Psychological intervention in women victims of childhood sexual abuse: a randomized controlled clinical trial comparing EMDR psychotherapy and trauma-focused cognitive behavioral therapy. Front Psychiatry. 2024 May 29;15:1360388. doi: 10.3389/fpsyt.2024.1360388. eCollection 2024. PMID 38868491

DOCUMENTS (1):
  • Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT04813224/ICF_000.pdf